CLINICAL TRIAL: NCT03951896
Title: Efficacy of Platelet Rich Plasma Injections in Patients With Adhesive Capsulitis of the Shoulder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Funda Atamaz Calis, Professor in Ege University School of Medicine, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP-AC
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Adhesive Capsulitis of Shoulder; Adhesive Capsulitis; Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The injection process was made with injectors coated with opaque adhesive tapes, and were prepared by another researcher who wasn't involved in injection or assessment. The statistical analyses were conducted without knowing the content of the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Experimental): Interventions:
  A venous blood sample of 8.5 ml were obtained from all patients. For the treatment group, the blood samples were treated with 1.5 ml ACD-A or sodium citrate to achieve anticoagulation. The blood was then centrifugated for 5 minutes with RCF 1200 G velocity to clump red blood cells, and then centrifugated for 10 minutes in same velocity to obtain platelet concentrate. 2 ml's of the resulting platelet rich plasma was injected to the shoulder of the subjects.
  Interventions: Biological: PRP
- Placebo (Placebo Comparator): For the control group, same amount of blood was sampled and they were given a same amount of waiting time with the other group, with the resulting injection preparate being 2 ml's of 0,9% saline instead.
  Interventions: Other: Saline injection

INTERVENTIONS:
Biological: PRP — A venous blood sample of 8.5 ml were obtained from all patients. For the treatment group, the blood samples were treated with 1.5 ml ACD-A or sodium citrate to achieve anticoagulation. The blood was then centrifugated for 5 minutes with RCF 1200 G velocity to clump red blood cells, and then centrifugated for 10 minutes in same velocity to obtain platelet concentrate. 2 ml's of the resulting platelet rich plasma was injected to the shoulder of the subjects.All of the injections were done every two weeks, for a total of 3 times using 21 G injection needles with injection technique of posterior approach.
  Other Names: Platelet Rich Plasma
  Arms: PRP
Other: Saline injection — 2 ml's of NaCl solution with 0,9% concentration was applied to the shoulders of the participants.
  Arms: Placebo

SUMMARY:
This study was done to investigate whether platelet rich plasma(PRP) injections are effective in the management of adhesive capsulitis of the shoulder(AC).Patients were randomized to 2 groups, and one group took PRP injections for 3 times every two weeks, while the other group took saline injections in same frequency and volume. A standardized exercise programme was also applied to all patients.

Patients were then evaluated with Shoulder Pain and Disability Index(SPADI), Visual analogous scales for pain and disability, Ranges of Movements and use of analgesics in before, after and 3rd month of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old and having a shoulder pain with restriction for 3 months at least, and 9 months at most(Pain VAS being >40 mm, and loss of ROM for affected side more than %25 of unaffected side).

Exclusion Criteria:

* Subjects were excluded if they had uncontrolled diabetes, active inflammatory diseases, ongoing pregnancy, severe anemia, psychiatric diseases that may affect compliance or cancer. Patients who had a history of trauma, recent injection therapies(<3 months), surgery or allergy to local anaesthetics, or signs of complex regional pain syndrome, local infections or use of non steroidal anti-inflammatory drugs throughout the study were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05-03 (Actual); Primary Completion 2015-09-04 (Actual); Study Completion 2015-09-04 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 3 months
  Shoulder Pain and Disability Index (SPADI) is a tool to assess pain and disability in patients with shoulder pain, which was extensively used in studies involving AC of the shoulder6, 15, 16. It consists of 5 questions in pain domain, and 8 questions in disability domain, which were expressed in a visual analogous scale.
Visual Analogous Scales for pain | 3 months
  Patients were asked to describe their pain, level of disability or treatment satisfaction on a 10 cm long line, with 0 point being "none", and 10 cm point being "highest possible". The proximity of the marked point to the 0 end was measured, and the results were recorded

SECONDARY OUTCOMES:
Visual Analogous Scales for disability | 3 months
  Patients were asked to describe their pain, level of disability or treatment satisfaction on a 10 cm long line, with 0 point being "none", and 10 cm point being "highest possible". The proximity of the marked point to the 0 end was measured, and the results were recorded
Shoulder ranges of motions | 3 months
  Shoulder range of motions were also evaluated at the time points that were mentioned, as secondary outcome measures. All of the measurements were done accordingly to the guidelines of American College of Orthopedic Surgeons by a conventional goniometer18, 19. The researcher who obtained the measurements was an experienced therapist in this field, and was blind to the treatment groups.
Analgesic use | 3 months
  Subjects were also asked about their needs of analgesic usage, namely acetaminophen. They were asked to write down each time they took an acetaminophen tablet of 500 mgs. The results were recorded as miligrams.

IPD SHARING:
Plan to Share IPD: No